CLINICAL TRIAL: NCT03285113
Title: A Single-arm, Open Label, Single Center Pilot Study to Confirm the Safety of Dorsal Root Ganglia (DRG) and Ultrahigh Frequency Spinal Cord Stimulator in Patients With Chronic Lower Limb Pain
Brief Title: A Study to Confirm the Safety of High Frequency DRG Stimulator in Patients With Chronic Lower Limb Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GiMer Medical (Industry)
Collaborators: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTC1601
Record Dates: First submitted 2017-09-14; First posted 2017-09-15 (Actual); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-12

CONDITIONS: Failed Back Surgery Syndrome; Complex Regional Pain Syndrome (CRPS)
MeSH Terms: conditions — Failed Back Surgery Syndrome; Complex Regional Pain Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrahigh Frequency Stimulation (Experimental): Patients with chronic lower limb pain will be treated with ultrahigh frequency stimulation via lead around DRG.
  Interventions: Device: GiMer Medical MN 1000 External Stimulator

INTERVENTIONS:
Device: GiMer Medical MN 1000 External Stimulator — Trial stimulator to generate pulsed ultrahigh frequency (>200KHz) electrical stimulation, delivered via lead around DRG, in treating pain. Similar with current market available Spinal Cord Stimulators but with a higher stimulation frequency (hundred KHz) range.

SUMMARY:
This study is a prospective, single-arm, open label, single center pilot study to confirm the safety of a ultrahigh frequency DRG stimulator in patients with chronic lower limb pain. The actual trial length is 5 days. Pts will be given ultrahigh frequency pulse stimulation, and VAS will be obtained after 3-4 hours of each stimulation.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, open label, single center pilot study to confirm the safety of a ultrahigh frequency DRG stimulator in patients with chronic lower limb pain. The actual trial length is 5 days. An initial eligibility screening within Day -14. Pt admitted to hospital on Day 1. The lead implantation is conducted on Day 2, and the 1st treatment starts after anesthesia recovery (Day 2 T1). If VAS >4 at 4 hours after the 1st treatment, the 2nd treatment will be conducted. VAS will be acquired 4 hours after the 2nd treatment. On Day 3, physical examination and vital signs will be collected. If VAS >4, the 3rd treatment will be provided. One hour after the 3rd treatment, the device will be removed and an X-ray will be taken. Three hours after the removal, VAS will be collected and then the patient will be discharged. VAS will be estimated by phone call on Day 4, and the patient will return to OPD for follow up examination on Day 5. The trial is completed on Day 5 visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≧20 and ≦75
2. Have a symptom of complex regional pain syndrome (CRPS), failed back surgery syndrome (FBSS), lower limb pain with or without lower back pain with a diagnosis related to spinal lesion and pain history of >6 months.
3. Have an average pain score >5 by Visual Analogue Scale (VAS) on inclusion.
4. Has failed to achieve adequate pain relief from prior pharmacologic treatments.
5. In the judgement of the investigator, the subject is an appropriate candidate for the trial procedure
6. The subject is willing and able to comply with the procedure and requirements of this trial.
7. The participant is able to understand and provide informed consent, and has signed their written informed consent in accordance with IRB requirements.

Exclusion Criteria:

1. Have evidence of a mental or psychological condition that affects pain perception and has difficulty/disability performing objective pain assessment, or have previously failed mental or psychological assessments administered by a psychiatrist that may be deemed to indicate the subject's lack of suitability for participation in this study.
2. Subject has exhibited escalating or changing pain condition within the past 30 days as evidenced by Investigator examination.
3. Be on anticoagulant medication with INR >1.5 or platelet count less than 100,000/μL, peripheral vascular diseases (PVDs), visceral pain or uncontrolled Diabetes mellitus (DM).
4. Has had corticosteroid therapy at an intended site of stimulation within the past 30 days.
5. Pain medication(s) dosages(s) are not stable for at least 30 days.
6. Has previously failed spinal cord stimulation therapy.
7. Currently has an active implantable device including ICD, pacemaker, spinal cord stimulator or intrathecal drug pump or subject requires magnetic resonance imaging (MRIs) or diathermy.
8. Has pain only within a cervical or thoracic distribution.
9. Have a current diagnosis of cancer with active symptoms
10. Have a known terminal illness with life expectancy less than one year
11. Have a systematic or local infection
12. Currently has an indwelling device that may pose an increased risk of infection.
13. Be pregnant or breast feeding
14. Have a medical history of drug or alcohol addiction within the past 2 years.
15. Participation in any investigational study in the last 30 days or current enrollment in any trial.
16. Be currently involved in an injury claim law suit or medically related litigation, including workers compensation.
17. Be a prisoner.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2018-02-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultrahigh Frequency Stimulation
Started | 10
Completed | 8
Not Completed | 2
Not completed — Unable to implant leads | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ultrahigh Frequency Stimulation
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety of Ultrahigh Frequency Treatment: Adverse Event (AE) and Serious AE (SAE)
Description: Number of Participants with Adverse Events and Serious Adverse Events
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrahigh Frequency Stimulation
Number analyzed (Participants) | 10
Participants | 5

2. Secondary Outcome: Change in Pain Measured by Visual Analog Scale (VAS)
Description: VAS: 0 (no pain) to 10 (max pain). Change in pain as a result of ultrahigh frequency DRG stimulation, as measured by VAS score compare to baseline VAS.
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ultrahigh Frequency Stimulation
Number analyzed (Participants) | 8
units on a scale | -2.7 (2.1)

3. Secondary Outcome: Incidence of Paresthesia
Description: If patients feel tingling during stimulation?
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrahigh Frequency Stimulation
Number analyzed (Participants) | 8
Participants | 0

4. Secondary Outcome: Change in Pain Medication Consumption
Description: Decrease in pain medication consumption, including Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) and weak opioids, compared to baseline
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrahigh Frequency Stimulation
Number analyzed (Participants) | 10
Participants | 3

ADVERSE EVENTS:
Time Frame: Trial duration (4 days)
Arm/Group | Ultrahigh Frequency Stimulation
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultrahigh Frequency Stimulation (N=10)
Incision site pain (Injury, poisoning and procedural complications) | 3 (3)
procedural headache (Injury, poisoning and procedural complications) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Increase blood pressure (Investigations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-02-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT03285113/Prot_000.pdf